CLINICAL TRIAL: NCT05618951
Title: Effects of Transverse Thoracic Mobilization With and Without Lower Trapezius Strengthening Exercises on Pain, Disability and Range of Motion in Patients With Mechanical Neck Pain
Brief Title: Effects of Transverse Thoracic Mobilization With and Without Lower Trapezius Strengthening Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/22/0153 Salba
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Mechanical Neck Pain
Keywords: Neck Pain; Trapezius muscle; Muscle strength; Range of Motion
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Lower Trapezius Strengthening Exercises (Experimental): Hot pack at neck area, upper trapezius stretching neck isometrics transverse mobilization glide and
  Lower Trapezius strengthening exercise includes:
  1. Latissimus pull down
  2. Prone V- raise
  3. Modified Prone Cobra and Standardized Physical Therapy treatment will be given as Hot pack at neck area, upper trapezius stretching, neck isometrics and transverse mobilization glide.
  Interventions: Other: Lower Trapezius Strengthening Exercises
- Group B: Standardized Physical Therapy (No Intervention): Hot pack at neck area, upper trapezius stretching neck isometrics transverse mobilization glide
  Group B given Standardized Physical therapy management

INTERVENTIONS:
Other: Lower Trapezius Strengthening Exercises — Lower Trapezius strengthening exercise includes:
  1. Latissimus pull down
  2. Prone V- raise
  3. Modified Prone Cobra
  Other Names: Standardized Physical Therapy
  Arms: Group A: Lower Trapezius Strengthening Exercises

SUMMARY:
Mechanical neck pain is a common musculoskeletal problem, worldwide. Patients with neck pain often have subjective complaints of muscle stiffness, tension, or tightness in addition to their pain located between the occiput and the third thoracic vertebra Approximately 68% of the total population has experienced neck pain at least once in their lifetime, and it easily transforms into a chronic state (that persists for more than 3 months). In today's society, this is conspicuous in many laborers due to the increased use of computers, where the neck and shoulders are maintained in static abnormal postures to look at the computer screens and become vulnerable to cause neck pain. The aim of the study is to determine the comparative effects of transverse thoracic mobilization with and without lower trapezius strengthening exercises on pain, disability and range of motion in patients with mechanical neck pain.

DETAILED DESCRIPTION:
A Randomized controlled trial will be conducted in physiotherapy outpatient department of Syed Medical Complex and Islam Hospital, Sialkot. Non-probability consecutive sampling will be used to collect the data. Sample size of 20 subjects with age group between 18 to 40 years will be taken. Data will be collected by using tools Numeric Pain Rate Scale (NPRS) for pain, Neck Disability Index (NDI) for disability and Universal Goniometer (UG) for range of motion of neck. An informed consent will be taken. A total of 20 subjects will be selected by following inclusion and exclusion criteria and will equally divided in to two groups by random number generator table. Both groups will come thrice per week for a total of 4 weeks. The data will be analyzed using SPSS software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the age range of 18-40 years with mechanical neck pain for at least 3months.
* Examination- Symptoms provoked by neck movement and/or palpation of neck musculature.
* Trapezius Strength Test -To assess lower trapezius muscle strength, patient in prone with shoulder 120 degree abducted and resist the shoulder extension diagonally.

Exclusion Criteria:

* Osteoporosis
* Tumors
* Vertebral fractures
* Diagnosed psychological disorders
* Neck pain associated with vertigo
* History of cervical and thoracic spine injury
* Cervical radiculopathy
* Traumatic neck injury
* Shoulder surgery

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rate Scale (NPRS) | follow up at 4th week
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults, including those with chronic pain. The NPRS is a segmented numeric version in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain.
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"). The NPRS takes <1 minute to complete The NPRS is a valid and reliable scale to measure pain intensity.
Universal Goniometer (UG) | follow up at 4th week
  A goniometer is an instrument that measures the available range of motion at a joint. To measure the range of motion physical therapists most commonly use a goniometer. It is necessary that a single notation system is used in goniometry. The neutral zero method (0 to 180- degree system) is the most widely used method. The same goniometer should always be used to reduce the chances of instrumental error.
Neck Disability Index (NDI) | follow up at 4th week
  This questionnaire has been designed to give information about neck pain and the ability to manage it in everyday life. Participants will answer every section and mark only the one box that applies in each section. If two or more statements are in any section related to the participant, mark only one box that is relevant closely. The questionnaire has 10 items concerning pain and activities of daily living, including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation. Each item is scored out of 5 (with the 'no disability' response given a score of 0), giving a total score of for the questionnaire 50. Higher scores represent more significant disabilities. The result can be expressed as a percentage or raw scores (out of 50).

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Mphil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Syed Medical Complex and Islam Hospital, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee KW, Kim WH. Effect of thoracic manipulation and deep craniocervical flexor training on pain, mobility, strength, and disability of the neck of patients with chronic nonspecific neck pain: a randomized clinical trial. J Phys Ther Sci. 2016 Jan;28(1):175-80. doi: 10.1589/jpts.28.175. Epub 2016 Jan 30. PMID 26957752
- [Background] Rodriguez-Sanz J, Malo-Urries M, Lucha-Lopez MO, Lopez-de-Celis C, Perez-Bellmunt A, Corral-de-Toro J, Hidalgo-Garcia C. Comparison of an exercise program with and without manual therapy for patients with chronic neck pain and upper cervical rotation restriction. Randomized controlled trial. PeerJ. 2021 Nov 24;9:e12546. doi: 10.7717/peerj.12546. eCollection 2021. PMID 34900443
- [Background] Wan-Hee Lee I-KC, Hye-Kang Park. The Effectiveness of Selective Lower Trapezius Strengthening Exercises on Pain, Muscle Function, and Scapular Position in Patients with Rounded Shoulder and Chronic Neck Pain. Physical Therapy Rehabilitation Science. 2021;10:503-11.
- [Background] Twinkle Y Dabholkar SY, Abichandani Deepa. Comparison of the efficacy of Maitland Thoracic Mobilization and Deep Neck Flexor Endurance Training Versus Only Deep Neck Flexor Endurance Training in Patients with Mechanical Neck Pain. Indian Journal of Physiotherapy and Occupational Therapy. 2014;8(3):6.
- [Background] Lee KS, Lee JH. Effect of maitland mobilization in cervical and thoracic spine and therapeutic exercise on functional impairment in individuals with chronic neck pain. J Phys Ther Sci. 2017 Mar;29(3):531-535. doi: 10.1589/jpts.29.531. Epub 2017 Mar 22. PMID 28356648
- [Background] Howell ER. The association between neck pain, the Neck Disability Index and cervical ranges of motion: a narrative review. J Can Chiropr Assoc. 2011 Sep;55(3):211-21. PMID 21886283
- [Background] Park SH, Lee MM. Effects of Lower Trapezius Strengthening Exercises on Pain, Dysfunction, Posture Alignment, Muscle Thickness and Contraction Rate in Patients with Neck Pain; Randomized Controlled Trial. Med Sci Monit. 2020 Mar 23;26:e920208. doi: 10.12659/MSM.920208. PMID 32202262
- [Background] Cunha AC, Burke TN, Franca FJ, Marques AP. Effect of global posture reeducation and of static stretching on pain, range of motion, and quality of life in women with chronic neck pain: a randomized clinical trial. Clinics (Sao Paulo). 2008 Dec;63(6):763-70. doi: 10.1590/s1807-59322008000600010. PMID 19060998
- [Background] Sowmya. Isometric Neck Exercises versus Dynamic Neck Exercises in Chronic Neck Pain. ournal of Nursing and Health Science. 2014;3(2):32-43.
- [Background] Behnoush B, Tavakoli N, Bazmi E, Nateghi Fard F, Pourgharib Shahi MH, Okazi A, Mokhtari T. Smartphone and Universal Goniometer for Measurement of Elbow Joint Motions: A Comparative Study. Asian J Sports Med. 2016 Jun 11;7(2):e30668. doi: 10.5812/asjsm.30668. eCollection 2016 Jun. PMID 27625754